CLINICAL TRIAL: NCT01624428
Title: Examining the Effects of Varenicline on Reward Responses,Cognition, and Tobacco Cues in Adolescent Smokers
Brief Title: Varenicline on Reward Responses and Cognition in Adolescent Smokers
Acronym: GRAND
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 1108008929
Record Dates: First submitted 2012-06-18; First posted 2012-06-20 (Estimated); Last update posted 2014-02-03 (Estimated); Status verified 2014-01

CONDITIONS: Tobacco Use Disorders
Keywords: Tobacco; Adolescent; Nicotine; Magnetic Resonance Imaging; Varenicline
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- varenicline (Active Comparator)
  Interventions: Drug: Varenicline
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Varenicline — 1 mg bid varenicline titrated over a 2 week period
  Other Names: Chantix
  Arms: varenicline
Drug: Placebo — 1 mg bid placebo titrated over a 2 week period
  Arms: Placebo

SUMMARY:
This is a pilot project using functional magnetic resonance imaging (fMRI) to examine the influence of varenicline on reward processing, cognitive control, and regulation of craving in adolescent smokers. We hypothesize that adolescent smokers receiving varenicline, when compared with those receiving placebo, will have differential brain responses to anticipation of rewards, during exposure to the Stroop task, and in response to tobacco cues.

DETAILED DESCRIPTION:
This is a pilot project using functional magnetic resonance imaging (fMRI) to examine the influence of varenicline on reward processing, cognitive control, and regulation of craving in adolescent smokers. We hypothesize that adolescent smokers receiving varenicline, when compared with those receiving placebo, will have increased activation of the ventral striatum (VS) in response to anticipation of rewards in the Monetary Incentive Delay Task (MIDT), decreased activation of the dorsolateral prefrontal cortex (dlPFC) during exposure to incongruent stimuli in the Stroop task, and reduced activation of the ventral striatum in response to tobacco cues, and increased activation of the dlPFC during regulation of responses to tobacco cues during the Regulation of Craving (ROC) task. The results of this pilot project will have important implications regarding the use of varenicline for treating tobacco dependence and understanding varenicline's neurobiological effects in adolescent smokers.

ELIGIBILITY:
Inclusion Criteria:

* Between 16-19 years of age
* Able to read and write English
* Smoking 5 or more cigarettes on a daily basis, for at least one year
* Not seeking smoking cessation treatment
* Weighing > 55 kg (121 lbs)

Exclusion Criteria:

* Current criteria for abuse or dependence on another psychoactive substance.
* Current diagnosis of any clinical significant psychiatric disease like major depressive disorder, panic or anxiety disorder, psychosis, schizophrenia, bipolar disorder.
* Those with a prior suicide attempt or with active suicidal ideation at baseline
* Any regular use of any psychoactive drugs including anxiolytics and antidepressants
* Pregnant or lactating girls: females of childbearing potential who are unwilling or unable to use an acceptable method of contraception from at least 14 days prior to study medication administration until 30 days after the last dose of study medication. Acceptable methods of contraception are: abstinence; any form of hormonal contraception such as Depo-Provera, daily oral contraceptive, transdermal patch, or Nuva-ring; intra-uterine device, sterilization; or double barrier contraception which is a combination of any two of the following methods: condoms, spermicide, diaphragm.
* Evidence or history of clinically significant neurological, hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, or allergic disease.
* History of prior use of or sensitivity to varenicline.
* Color-blindness
* History of significant head trauma
* Metal in body
* Other medical conditions contra-indicated for MRI
* Past history of marked irritability or agitation when attempting to quit smoking, determined by the Minnesota Nicotine Withdrawal Questionnaire.

Ages: 16 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2012-06; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
neural responses to the MIDT | During MRI following14 days of varenicline treatment
  The Monetary Incentive Delay Task (MIDT) will be administered during the fMRI at the end of 14 days of varenicline treatment
neural responses to the ROC | During MRI following14 days of varenicline treatment
  The Regulation of Craving (ROC)will be administered during the fMRI at the end of 14 days of varenicline treatment
neural responses to the Stroop | During MRI following14 days of varenicline treatment
  The Stroop will be administered during the fMRI at the end of 14 days of varenicline treatment

CONTACTS AND LOCATIONS:
Overall Officials: Suchitra Krishnan-Sarin, Ph.D., Principal Investigator — Yale University
Locations (1):
- Substance Abuse Center, New Haven, Connecticut, United States